CLINICAL TRIAL: NCT02103205
Title: Effect of Infant Formula With Bovine Lactoferrin and Low Iron Concentration on Infant Health and Immune Function
Acronym: LIME
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: University of California (Other); Mead Johnson Nutrition (Industry)
Responsible Party: Principal Investigator, Staffan Berglund, MD, PhD, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LIME2014
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Health of Formula-fed Children; Infant Infections in Formula-fed Children; Iron Status of Formula-fed Children
Keywords: Lactoferrin; Infant formula; Iron
MeSH Terms: interventions — Food, Formulated; Lactoferrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low iron, with lactoferrin (Active Comparator): Low iron, with lactoferrin
  Interventions: Dietary Supplement: Formula with low iron concentration (2 mg/L) supplemented with bovine lactoferrin
- Low iron, no lactoferrin (Active Comparator): Low iron, no lactoferrin
  Interventions: Dietary Supplement: Formula with low iron concentration (2mg/L) without lactoferrin
- Normal iron, no lactoferrin (Placebo Comparator): Normal iron, no lactoferrin
  Interventions: Dietary Supplement: Formula with normal iron concentration (8 mg/L) without lactoferrin

INTERVENTIONS:
Dietary Supplement: Formula with low iron concentration (2 mg/L) supplemented with bovine lactoferrin
  Arms: Low iron, with lactoferrin
Dietary Supplement: Formula with low iron concentration (2mg/L) without lactoferrin
  Arms: Low iron, no lactoferrin
Dietary Supplement: Formula with normal iron concentration (8 mg/L) without lactoferrin
  Arms: Normal iron, no lactoferrin

SUMMARY:
Breast milk is the gold standard of early infant nutrition and breastfed infants have advantages in several short and long term outcomes compared to those formula-fed.

The first aim of this study is to evaluate the effect of adding bovine lactoferrin to infant formula. The general hypothesis is that bovine lactoferrin reduces some of the previously observed differences between formula-fed and breast-fed infants with regard to health and development. The main outcome studied is the effect on immune function. The second aim is to study the effects of lower iron concentration in infant formula and to test the hypothesis that iron can be lowered without negative effects on health and development. The main outcome studied here is iron status. Other outcomes in this trial are microbiota composition, metabolomics, growth, body composition and cognitive development.

To test the lactoferrin hypothesis, formula-fed infants will be recruited and fed a low iron (2 mg/L) control formula, or the same formula supplemented with bovine lactoferrin. To test the iron hypothesis, a third group will be fed the same formula (no lactoferrin) with higher iron concentration (8 mg/L). Group allocation for all formula-fed infants will be double-blind randomized. Additionally, breast-fed infants will be recruited and used as a reference group (gold standard).

ELIGIBILITY:
Inclusion Criteria:

Formula-fed healthy infants at 6 +/- 2 weeks of age with:

* birth weight 2500-4500 g
* gestational age at birth ≥ 37 completed weeks
* no chronic disease or neonatal diagnoses believed to affect any outcome
* no given blood transfusions or iron supplements

Exclusion Criteria:

-

Ages: 4 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 252 (Actual)
Dates: Start 2014-06; Primary Completion 2019-05 (Actual); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of infections | Up to 12 months of age
  Morbidity journal, Health questionnaire
Cytokine levels | At 6 months of age
  IL-2, TNF-alpha
Iron status | At 6 months of age
  s-ferritin, s-transferrin, s-iron, s-transferrin receptor concentration, reticulocyte Hb

SECONDARY OUTCOMES:
Dietary intake | At baseline, 3, 4, 5, 6 and 12 months of age
  Dietary journal
Growth | At baseline, 4, 6, 12 months of age and 6 years of age
  Anthropometric data, Body Composition (PeaPod)
Bloodpressure | At baseline, 4, 6, 12 months of age and 6 years of age
Antibody response to vaccines | At baseline, 4, 6 and 12 months of age
  s-levels of specific antibodies to vaccines (DTP, Hib, PC)
Gut microbiota | At baseline, 4, 6, 12 months of age and 6 years of age
  Stool samples
Saliva proteins | At 4 months of age
  Saliva total protein content, lactoferrin, saliva-peroxidase, IgA and amylase
Inflammatory markers | At baseline, 4, 6 and 12 months of age and 6 years age
  s-hsCRP, s-calprotectin
Cognitive development and behavior | At 1 and 6 years of age
  Bayley III, Wechsler Intelligence Scale for Children (WISC), Behavioral questionnaire
s-hepcidin | At baseline, 4, 6, 12 months of age and 6 years of age
Metabolomics | At baseline, 4, 6, 12 months of age and 6 years of age
  Analyzed in urine and serum samples
Amino acids | At 4 and 6 months of age
  p-amino acids
Blood urea nitrogen | At 4 and 6 months of age
  p-urea nitrogen
Cytokine levels | At baseline, 4, 6, 12 months of age and 6 years of age
  IL-2 and TNF alpha at baseline, 4 and 12 months of age and 6 years of age. Six additional cytokines at baseline, 4, 6 and 12 months of age and 6 years of age.
Iron status | At baseline, 4 and 12 months of age and 6 years of age
  s-ferritin, s-transferrin, s-iron, s-transferrin saturation, s-transferrin receptor concentration, retuiculocyte Hb

OTHER OUTCOMES:
Lactoferrin in breastmilk | At baseline, 4 and 6 months of age
  Analyzed from mothers to the control group of breast fed infants.

CONTACTS AND LOCATIONS:
Overall Officials: Staffan K Berglund, MD, PhD, Principal Investigator — Umeå University; Olle Hernell, Professor, Principal Investigator — Umeå University; Bo Lönnerdal, Professor, Principal Investigator — University of California; Carolyn Slupsky, PhD, Principal Investigator — University of California
Locations (1):
- Umeå University, Department of Clinical Sciences, Umeå, Sweden

REFERENCES:
- [Derived] Bjormsjo M, Hernell O, Lonnerdal B, Berglund SK. Immunological Effects of Adding Bovine Lactoferrin and Reducing Iron in Infant Formula: A Randomized Controlled Trial. J Pediatr Gastroenterol Nutr. 2022 Mar 1;74(3):e65-e72. doi: 10.1097/MPG.0000000000003367. PMID 34908015